CLINICAL TRIAL: NCT06435728
Title: Predictive Value of Combining Angio-Based Index of Microcirculatory Resistance and Fractional Flow Reserve in Patients With STEMI
Brief Title: Predictive Value of Combining AccuIMR and AccuFFR in Patients With STEMI
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: D2023173
Record Dates: First submitted 2024-05-26; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction; Prognosis
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI: Patients with STEMI who underwent primary PCI and were hospitalized at Peking University Third Hospital between January 2017 and March 2022
  Interventions: Diagnostic Test: AccuIMR and AccuFFR

INTERVENTIONS:
Diagnostic Test: AccuIMR and AccuFFR — AccuFFR and AccuIMR were obtained by reviewing coronary angiography at the time of primary PCI

SUMMARY:
Patients with acute myocardial infarction were enrolled retrospectively. The fractional flow reserve (AccuFFR) and microcirculatory resistance index (AccuIMR) based on coronary angiography were analyzed, and the relationship between FFR and IMR and the prognosis of patients with acute myocardial infarction was analyzed

DETAILED DESCRIPTION:
We retrospectively enrolled STEMI patients who underwent PCI in Peking University Third Hospital. The fractional flow reserve (AccuFFR) and microcirculatory resistance index (AccuIMR) based on coronary angiography were obtained by analyzing the coronary angiography images. The prognosis of patients was obtained by searching inpatient and outpatient systems and telephone follow-up. The relationship between AccuFFR, AccuIMR and prognosis was statistically analyzed

ELIGIBILITY:
Inclusion Criteria:

* Age of >18 years;
* Onset-to-treatment time of ≤12 h, meeting the diagnostic criteria for STEMI;
* underwent primary PCI within 12 h of symptom onset and achieved successful PCI in the culprit vessel;
* Availability of complete clinical data

Exclusion Criteria:

* severe tortuosity and overlap of the target vessel;
* poor-quality coronary angiography images;
* missing two coronary angiography images >25° apart

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI who underwent primary PCI and were hospitalized at Peking University Third Hospital between January 2017 and March 2022.
Sampling Method: Non-Probability Sample
Enrollment: 1297 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
MACE | 3 years after myocardial infarction
  cardiovascular death, all-cause death, readmission for heart failure (HF), and recurrent coronary events

SECONDARY OUTCOMES:
recurrent coronary events | 3 years after myocardial infarction
  nonfatal myocardial infarction, unplanned PCI, and unplanned coronary artery bypass grafting

CONTACTS AND LOCATIONS:
Overall Officials: Ming Cui, Dorctor, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Xie P, Hu Y, Zhou Y, Zhao W, Xu X, Zhu D, Mi L, Xiang J, Cui M. Predictive Value of Combining Angio-Based Index of Microcirculatory Resistance and Fractional Flow Reserve in Patients with STEMI. Can J Cardiol. 2025 Jul;41(7):1363-1371. doi: 10.1016/j.cjca.2025.02.003. Epub 2025 Feb 6. PMID 39922306